CLINICAL TRIAL: NCT04338438
Title: Apatinib Plus S-1 for Advanced Gastric Cancer Refractory to Oxaliplatin Plus Capecitabine Combination Therapy: A Single-arm, Phase-2, Home-based Trial
Brief Title: Efficacy and Safety of Apatinib Combined With S-1 for Patients With Advance Gastric Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Zhongtao Zhang, Professor, Beijing Friendship Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BFH-Apatinib&S-1
Record Dates: First submitted 2020-04-05; First posted 2020-04-08 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Gastric Cancer
Keywords: late-stage
MeSH Terms: conditions — Stomach Neoplasms | interventions — apatinib; S 1 (combination)

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Apatinib Mesylate tablets combined with S-1 capsules (Experimental): single arm trial: apatinib 500 mg once daily, across entire cycle and S-1 60 mg twice daily, on the first 14 days of a 21-day cycle. Medication was continued until the disease progression, withdrawal requirement, or intolerable adverse events
  Interventions: Drug: Apatinib Mesylate tablets combined with S-1 capsules

INTERVENTIONS:
Drug: Apatinib Mesylate tablets combined with S-1 capsules — Apatinib Mesylate tablets combined with S-1 capsules, p.o.

SUMMARY:
This is a single-arm, interventional study aimed to observe the efficacy and safety of Apatinib combined with S-1 for patients with advanced gastric cancer refractory to oxaliplatin plus capecitabine combination therapy

ELIGIBILITY:
Inclusion Criteria Each patient must meet the following criteria to be enrolled in this study.

* The patient has provided signed informed consent and is amenable to compliance with protocol schedules and testing.
* The patient is at least 18 years of age (or of an acceptable age according to local regulations, whichever is older).
* The patient has an Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 -2 at study entry.
* The patient has a histopathologically or cytologically confirmed diagnosis of gastric or gastroesophageal junction (GEJ) adenocarcinoma.
* The patient has metastatic disease or locally advanced, unresectable or recurrent disease.
* The patient has experienced documented objective radiographic or clinical disease progression (eg, any new or worsening malignant effusion documented by ultrasound examination) which may be confirmed by pathologic criteria (histology and/or cytology) if appropriate, during first-line therapy, or within 6 months after the last dose of first-line therapy with Oxaliplatin plus Capecitabine doublet with or without anthracycline (epirubicin or doxorubicin) for unresectable or metastatic disease.
* The patient has resolution to Grade ≤1 by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE), Version 4.03, of all clinically significant toxic effects of prior locoregional therapy, surgery, or other anticancer therapy.
* The patient has adequate organ function, defined as:

  1. Total bilirubin ≤1.5 times upper limit of normal value (ULN), aspartate transaminase (AST) and alanine transaminase (ALT) ≤3 ULN for ALT/AST if no liver metastases, <5 ULN if liver metastases;
  2. Serum creatinine ≤1.5 ULN or calculated creatinine clearance (per the Cockcroft-Gault formula or equivalent and/or 24-hour urine collection) ≥50 mL/min;
  3. Absolute neutrophil count (ANC) ≥1.5 109 /L, hemoglobin ≥ 9 g/dL (5.58 mmol/L; packed red blood cell transfusions are not allowed within one week prior to baseline hematology profile), and platelets ≥100 109 /L;
  4. International Normalized Ratio (INR) ≤ 1.5 or Prothrombin time (PT) ≤1.5 ULN;
  5. Partial thromboplastin time (PTT/APTT) ≤ 1.5 ULN.
* The patient's urinary protein is ≤1+ on dipstick or routine urinalysis. If urine dipstick or routine analysis indicates proteinuria ≥2+, then a 24-hour urine must be collected and must demonstrate <1000 mg of protein in 24 hours to allow participation in the study.
* The patient, if female, is surgically sterile, postmenopausal, or compliant with a highly effective contraceptive method (failure rate <1%) during and for 12 weeks after the treatment period (oral hormonal contraception alone is not considered highly effective and must be used in combination with a barrier method). If male, the patient is surgically sterile or compliant with a highly effective contraceptive regimen during and for 6 months after the treatment period. The label requirements with regard to the methods and duration of contraception during and after treatment with paclitaxel can differ between countries. Country specific requirements will apply only if they are more stringent than those already stipulated in the protocol.

Exclusion Criteria Patients who meet any of the following criteria will be excluded from the study.

* The patient has squamous cell or undifferentiated gastric cancer.
* The patient has undergone major surgery within 28 days prior to medications, or central venous access device placement within 7 days prior to medications.
* The patient has received any chemotherapy other than Oxaliplatin plus Capecitabine for advanced gastric or GEJ adenocarcinoma.
* The patient has received previous systemic chemotherapy with a cumulative dose of >900 mg/m2 of epirubicin or >400 mg/m2 of doxorubicin.
* The patient has received any previous systemic therapy (including investigational agents) targeting vascular endothelial growth factor(VEGF) or the vascular endothelial growth factor receptor(VEGFR) signaling pathways. Other previous targeted therapies are permitted, if stopped at least 28 days prior to randomization.
* The patient has a history of deep vein thrombosis, pulmonary embolism, or any other significant thromboembolism (venous port or catheter thrombosis or superficial venous thrombosis are not considered "significant") during the 3 months prior to randomization.
* The patient is receiving therapeutic anticoagulation with warfarin, low-molecular weight heparin or similar agents. Patients receiving prophylactic, low-dose anticoagulation therapy are eligible provided that the coagulation parameters defined in the inclusion criteria (INR ≤1.5 and PTT/APTT ≤1.5 ULN) or (PT ≤1.5 ULN and PTT/aPTT ≤1.5 ULN) are met.
* The patient is receiving chronic therapy with nonsteroidal anti-inflammatory agents (NSAIDs, eg, indomethacin, ibuprofen, naproxen or similar agents) or other anti-platelet agents (eg, clopidogrel, ticlopidine, dipyridamole, anagrelide). Aspirin use at doses up to 325 mg/day is permitted.
* The patient has significant bleeding disorders, vasculitis, or had a significant bleeding episode from the gastrointestinal tract within 3 months prior to study entry.
* History of gastrointestinal perforation and/or fistulae within 6 months prior to medications.
* The patient has symptomatic congestive heart failure (New York Heart Association II-IV) or symptomatic or poorly controlled cardiac arrhythmia.
* The patient has experienced any arterial thrombotic event, including myocardial infarction, unstable angina, cerebrovascular accident, or transient ischemic attack, within 6 months prior to randomization.
* The patient has uncontrolled arterial hypertension ≥150/≥90 mm Hg despite standard medical management.
* The patient has a serious or non healing wound or peptic ulcer or bone fracture within 28 days prior to medications.
* The patient has a bowel obstruction, history or presence of inflammatory enteropathy or extensive intestinal resection (hemicolectomy or extensive small intestine resection with chronic diarrhea), Crohn's disease, ulcerative colitis, or chronic diarrhea.
* The patient has a serious illness or medical condition(s) including, but not limited to the following:

  1. Known human immunodeficiency virus infection or acquired immunodeficiency syndrome-related illness;
  2. Active or uncontrolled clinically serious infection;
  3. Previous or concurrent malignancy except for basal or squamous cell skin cancer and/or in situ carcinoma of the cervix, or other solid tumors treated curatively and without evidence of recurrence for at least 3 years prior to the study;
  4. Uncontrolled metabolic disorders or other nonmalignant organ or systemic diseases or secondary effects of cancer that induce a high medical risk and/or make assessment of survival uncertain;
  5. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the Investigator would make the patient ineligible for entry into this study;
  6. History or evidence of known central nervous system metastases or carcinomatous meningitis;
  7. Known allergy or hypersensitivity to monoclonal antibody treatment or any components used in the apatinib;
  8. Known allergy or hypersensitivity to S-1 or any components used in the S-1 preparation.
* The patient is pregnant or breastfeeding.
* The patient is currently enrolled in, or discontinued within the last 28 days from a clinical trial involving an investigational product or non-approved use of a drug, or concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study. Patients participating in surveys or observational studies are eligible to participate in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
median progression-free survival(mPFS) | 2 years
  The median duration of time between when a patient with oncological disease receives treatment and when the disease progresses or death due to any cause occurs.
median overall survival(mOS） | 2 years
  The median time from treatment to the last follow-up or death.

SECONDARY OUTCOMES:
objective response rate(ORR) | 2 years
  The rate of patients achieved complete response or partial response
disease control rate(DCR) DCR | 2 years
  The rate of patients achieved complete response or partial response or solid disease.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Deng, M.D., Study Director — Beijing Friendship Hospital

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 2020.12~
Access Criteria: via reasonable email requests

REFERENCES:
- [Background] Noh SH, Park SR, Yang HK, Chung HC, Chung IJ, Kim SW, Kim HH, Choi JH, Kim HK, Yu W, Lee JI, Shin DB, Ji J, Chen JS, Lim Y, Ha S, Bang YJ; CLASSIC trial investigators. Adjuvant capecitabine plus oxaliplatin for gastric cancer after D2 gastrectomy (CLASSIC): 5-year follow-up of an open-label, randomised phase 3 trial. Lancet Oncol. 2014 Nov;15(12):1389-96. doi: 10.1016/S1470-2045(14)70473-5. Epub 2014 Oct 15. PMID 25439693
- [Background] Sakuramoto S, Sasako M, Yamaguchi T, Kinoshita T, Fujii M, Nashimoto A, Furukawa H, Nakajima T, Ohashi Y, Imamura H, Higashino M, Yamamura Y, Kurita A, Arai K; ACTS-GC Group. Adjuvant chemotherapy for gastric cancer with S-1, an oral fluoropyrimidine. N Engl J Med. 2007 Nov 1;357(18):1810-20. doi: 10.1056/NEJMoa072252. PMID 17978289
- [Background] Lan CY, Wang Y, Xiong Y, Li JD, Shen JX, Li YF, Zheng M, Zhang YN, Feng YL, Liu Q, Huang HQ, Huang X. Apatinib combined with oral etoposide in patients with platinum-resistant or platinum-refractory ovarian cancer (AEROC): a phase 2, single-arm, prospective study. Lancet Oncol. 2018 Sep;19(9):1239-1246. doi: 10.1016/S1470-2045(18)30349-8. Epub 2018 Aug 3. PMID 30082170
- [Background] Li J, Qin S, Xu J, Guo W, Xiong J, Bai Y, Sun G, Yang Y, Wang L, Xu N, Cheng Y, Wang Z, Zheng L, Tao M, Zhu X, Ji D, Liu X, Yu H. Apatinib for chemotherapy-refractory advanced metastatic gastric cancer: results from a randomized, placebo-controlled, parallel-arm, phase II trial. J Clin Oncol. 2013 Sep 10;31(26):3219-25. doi: 10.1200/JCO.2013.48.8585. Epub 2013 Aug 5. PMID 23918952
- [Background] Roviello G, Ravelli A, Polom K, Petrioli R, Marano L, Marrelli D, Roviello F, Generali D. Apatinib: A novel receptor tyrosine kinase inhibitor for the treatment of gastric cancer. Cancer Lett. 2016 Mar 28;372(2):187-91. doi: 10.1016/j.canlet.2016.01.014. Epub 2016 Jan 18. PMID 26797419
- [Background] Liang W, Guan W, Chen R, Wang W, Li J, Xu K, Li C, Ai Q, Lu W, Liang H, Li S, He J. Cancer patients in SARS-CoV-2 infection: a nationwide analysis in China. Lancet Oncol. 2020 Mar;21(3):335-337. doi: 10.1016/S1470-2045(20)30096-6. Epub 2020 Feb 14. No abstract available. PMID 32066541
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2020. CA Cancer J Clin. 2020 Jan;70(1):7-30. doi: 10.3322/caac.21590. Epub 2020 Jan 8. PMID 31912902
- [Background] Zong L, Abe M, Seto Y, Ji J. The challenge of screening for early gastric cancer in China. Lancet. 2016 Nov 26;388(10060):2606. doi: 10.1016/S0140-6736(16)32226-7. No abstract available. PMID 27894662
- [Derived] Jing C, Bai Z, Zhang J, Jiang H, Yang X, Yan S, Yin J, Cai J, Zhang Z, Deng W. Apatinib plus S-1 for previously treated, advanced gastric or gastro-oesophageal junction adenocarcinoma: a phase 2, single-arm, prospective study. J Gastrointest Oncol. 2021 Oct;12(5):2035-2044. doi: 10.21037/jgo-21-186. PMID 34790371